CLINICAL TRIAL: NCT04272970
Title: Characterization of New Candidate Genes in Cases of Human Inherited Thrombocytopenia (CATCH). Molecular Etiologies in Cases of Thrombocytopenia
Brief Title: Characterization of New Candidate Genes in Cases of Human Inherited Thrombocytopenia (CATCH)
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: C19-08; 2019-A01351-56 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-01-21; First posted 2020-02-17 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Thrombocytopenia; Inherited Platelet Disorder
Keywords: Familial thrombocytopenia; Molecular etiology
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: Within each family that will be studied for functional studies of platelets and MKs, subjects both harboring a variant gene / protein and presenting with CT will be compared to non CT family members with a normal gene / protein (control subjects) in parallel investigation ; when family control subject(s) will not be available, a subject external to the family with no evidence for CT will be recruited as a control subject
Who Masked: Participant
Masking Description: Each participant will receive at the time of recruitment a normalized code number that will remain confidential for the investigators, and which will hide his / her full identity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New gene / protein variant functional study (Active Comparator): Morphological and functional studies of circulating blood platelets and hematopoietic progenitor cells, in order to prove the pathogenicity of variants of new genes potentially involved in constitutional familial thrombocytopenia.
  Interventions: Diagnostic Test: Validation of a new gene / protein variant implicated in familial CT
- Normal gene / protein variant functional study (Sham Comparator): Morphological and functional studies of circulating blood platelets and hematopoietic progenitor cells, in order to provide control observations / analyses / measures for the "Active Comparator" arm
  Interventions: Diagnostic Test: Validation of a new gene / protein variant implicated in familial CT

INTERVENTIONS:
Diagnostic Test: Validation of a new gene / protein variant implicated in familial CT — Realize a blood sample to perform functional studies of circulating blood platelets and hematopoietic progenitor cells, in order to prove the pathogenicity of variants of new genes potentially involved in constitutional thrombocytopenia.

SUMMARY:
Circulating blood platelets are small cellular elements that help to control bleeding (a process called hemostasis) and to avoid hemorrhage when blood vessels are injured. Platelets originate from cells in the bone marrow, the megakaryocytes (MKs), following a complex process of morphological transformation and maturation, which finally leads to the production of blood platelets. Multiple genes are implicated in this process. Constitutive thrombocytopenia (CT) are rare hematological diseases characterized by a decreased number of circulating platelets that are often larger than normal, that may lead to more or less severe hemorrhagic events. However, CT can be difficult to diagnose and differentiate from various forms of acquired thrombocytopenia. The ultimate diagnosis for CT is thus based on the molecular diagnosis, obtained by identifying and characterizing the abnormal gene and protein. About 40 genes / proteins have been identified so far as causal in CT, however, in about half of the patients suspected to have CT, genomic analysis does not detect a variant in one of these genes, and etiology of CT thus remains unknown. But insuring the diagnosis of CT is important: it will avoid misdiagnosis and inefficient or deleterious therapeutic interventions, while allowing a proposal of an adapted curative/preventive medical action. At the Resource and Competence Center for Constitutional Hemorrhagic Diseases (CRCMHC) (University Hospital Robert Debré, Paris, France), the investigating team has evidenced in unrelated patients presenting with familial forms of thrombocytopenia and no known molecular diagnosis, variants of genes not yet described as formally implicated in the occurrence of CT. Molecular genetic evidence must be completed by functional studies. Such functional studies are conducted in a research laboratory from the National Institute for Health and Medical Research (Inserm), "Innovative Therapies in Haemostasis (IThEM)" (Faculty of Medical Sciences, University of Paris, Paris, France), and include:

* an evaluation of how blood progenitor cells mature into MKs, by comparing cells obtained from patients to those of members free of the disease (the latter taken as normal control subjects);
* an evaluation of platelet functionalities, such as ability to form a blood clot similar to what happens during hemostasis, with the aim to detect not only quantitative (number and size) but also any qualitative (functions) defects;
* an evaluation of the ultrastructure (the structure of intracellular components) and biochemistry of MKs and platelets, focusing on the molecular pathways the variant protein is implicated in.

This clinical trial is aimed to precisely delineate the mechanism of action of newly identified CT genetic variants, and will fulfill the aims of (1) offering the patient(s) a formal molecular diagnosis of CT, (2) ameliorating patients' medical support, both for diagnosis and therapy, (3) providing patients and family members with a pertinent genetic counseling, and (4) expanding the validated panel of genes implicated in CT to be explored in new suspected cases of CT. It will also help in extending the basic knowledge of the process of MK and platelet formation.

DETAILED DESCRIPTION:
Circulating blood platelets are essential in the maintenance of vascular integrity and functionality in numerous pathophysiological situations, such as the control of hemorrhagic or thrombotic events. Platelets are released into the circulation from highly specialized bone marrow cells, the megakaryocytes (MKs) that undergo a complex process of differentiation and maturation. This process starts with the differentiation of bone marrow hematopoietic progenitor cells (HPC) into enlarging, polyploid immature MKs that evolve into giant cells apposed on the bone marrow microvasculature, and finally release into the blood stream fragments of their cytoplasm that make the circulating platelets. This ultimate step of MK maturation is called thrombopoiesis. Multiple genes are implicated in the whole process, and particularly in precisely defining both the size and number of circulating platelets. Constitutive thrombocytopenia (CT) are rare hematological diseases etiologically heterogeneous, characterized by a markedly decreased number of circulating platelets. In most of the cases, thrombocytopenia is accompanied by a change in cell size that very often appears as an increased mean volume. Thrombocytopenia is a life-long status for the patient, and when circulating platelets are strongly diminished, this may lead to hemorrhagic events of variable severity that may require urgent intervention such as transfusion of blood products. Depending on the gene that is altered, CT may be present in parallel with other blood cell diseases, such myelodysplastic syndrome or leukemia, or even with extra-hematological syndromes, such nephropathy, deafness, etc. However, CT can be difficult to diagnose and difficult to differentiate from various forms of acquired thrombocytopenia, such as idiopathic or drug-induced thrombocytopenia. The ultimate diagnosis for CT is based on the molecular diagnosis that must show that a variant gene and protein harboring identified mutation(s) do alter platelet production and result in clinical CT.

Knowledge about the genetic basis of CT is continuously expanding, with ~ 40 genes identified so far as causative in CT cases. This identification is based on rigorous criteria such as (1) bioinformatics-based evaluation of the pathogenicity of the mutations, (2) genotype - phenotype association in informative CT families, and (3) reproduction of the molecular and cellular abnormalities noted in the patients by using experimental cellular or animal models. All implicated genes and proteins act at important steps during MK differentiation / maturation, and particularly during thrombopoiesis. In addition to important biomedical outcomes, characterization of mutations of these genes and the impact they have on various biological processes is also an irreplaceable source of discoveries in basic cell biology. However, in about half of clinically suspected CT cases, genomic analysis of the known implicated genes does not recover a variant in one of these genes. Thus, some etiologies of CT are yet unknown, and there is still a lot of investigation to perform in order to expand and complement the list of genes and mutations implicated in CT. This is important for the patients and families, because insuring the diagnosis of CT will avoid misdiagnosis and its potential inefficient or deleterious therapeutic interventions, including blood products transfusion when non pertinent, while allowing a proposal of an adapted curative/preventive medical action, especially when the CT is associated with an extra-platelet or extra-hematological syndrome.

At the Resource and Competence Center for Constitutional Hemorrhagic Diseases (CRCMHC; University Hospital Robert Debré, Paris, France), the investigating team has built a cohort of more than 650 subjects presenting with CT, which only about half have received a genetic diagnosis. Among the patients without such a molecular diagnosis, several, unrelated patients with a familial form of thrombocytopenia have been recently investigated by the investigating team and shown to harbor variants of genes not yet described as formally implicated in the occurrence of CT. However, clinical and molecular genetic evidence must be completed by functional studies of the corresponding variant proteins in their cellular environment, and this experimental, cell biology approach of the CT pathology makes the basis of the present clinical trial. Such functional studies will include:

* an evaluation of how blood HPC obtained from patients and family members either with CT or free of the disease (the latter taken as normal control subjects), differentiate into MKs when seeded in culture dishes, then mature into MKs forming proplatelets, that are similar to the early platelets formed in the bone marrow before their release into blood. The purpose is to observe and analyze any morphological and protein expression abnormality that may be present in CT cells, and absent in non-CT cells. The techniques used are cell culture, microscope observation and analysis, both qualitative and quantitative, of modifications in protein expression and / or distribution in cells, using probes such as antibodies raised against the proteins of interest;
* an evaluation of platelet functionalities, such as their ability to adhere to the surface of a blood vessel, then to aggregate, an hallmark of their essential role in stopping bleeding, and to retract a clot, characteristic of their role in the sealing of a damaged blood vessel, thereby avoiding infections and preparing the tissue for repair. The aim here is to observe and analyze any alteration of these highly platelet-specific functions during hemostasis in CT platelets compared to normal platelets, because certain genes affecting the platelet production in the bone marrow may also play a role in the functions of circulating platelets. Techniques to be used are microscopy imaging of platelet adherence to experimental protein-coated surfaces, or to genuine vascular material;
* an evaluation of the MK/platelet ultrastructure and biochemistry, focusing on the intracellular molecular pathways the variant protein is implicated in. Techniques to use for this purpose are confocal or electronic microscopy, protein extraction, purification and analysis.

These experimental studies are conducted in a research laboratory from the National Institute for Health and Medical Research (Inserm), "Innovative Therapies in Haemostasis (IThEM)" (Faculty of Pharmacy - University of Paris, Paris, France). The laboratory is acting in this clinical trial on a collaborative basis with the CRCMHC, which is operating upstream for the medical, clinical and genetic characterization of patients and family members who may be then asked for enrollment in the trial. The IThEM laboratory has also the expertise to generate cellular models for the study of one particular gene and protein variant, that can be experimentally introduced into laboratory human primary cells or cell lines in order to reproduce the biologic alterations originally observed in cells from the CT patients. This serves to strengthen the demonstration that the variant gene is truly pathogenic, but this part of the study is outside the present clinical trial because it does not require access to biological material from the patients and family members in order to be performed.

In the whole, this clinical trial is aimed to precisely delineate the mechanism of action at the molecular and cellular levels of newly identified CT-associated gene variants, in order to confirm or, conversely, invalidate the pathogenicity of the variant gene. It will fulfill several objectives, (1) to offer the patient(s) a formal molecular diagnosis of CT, (2) to precise and elucidate the phenotypic presentation of the form of CT generated by this variant, (3) to help to ameliorate patients' medical support, both for diagnosis and therapy, particularly if CT have extra-platelet and / or extra-hematological counterparts, (4) to provide patients and family members a pertinent genetic counseling, and (5) to expand the validated panel of genes implicated in CT and to be explored on presentation of a new suspected case of CT. It will also help in extending the basic knowledge of the process of megakaryocytopoiesis and thrombopoiesis, both normal and pathological.

ELIGIBILITY:
Inclusion Criteria:

* platelet count < 150.000/µl for at least 6 months
* thrombocytopenia in at least one family member
* weight > 35 kg
* no pathogenic variant (already reported or suspected) in genes causative for inherited CT
* harboring a variant potentially pathogenic in a gene potentially implicated in the megakaryopoiesis or platelet production, this variant being harbored also by the affected family members, and not by the non-affected family members .

Exclusion Criteria:

* Pregnant woman
* Subject with an anemia: Hb < 8g/dl
* Subject with a behavior disorder
* Subject with a hemostasis disease added (Willebrand disease, hemophilia, ...)
* Subject with another suspected cause of thrombopenia (drug, infection, ...)
* Subject taking a drug interfering on the platelet production
* Subject protected by a legal measure
* Subject participating to another program research, leading to larger blood volume than authorized

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Validation of new genes potentially involved in the occurrence of CT by determination of the amount of the protein produced and its effect on the megakaryocytes producing platelets aspect in culture | 6 months
  Functional study of variants altering these new genes, identified in patients and their family members presenting a CT. This study will include the determination of the amount of the protein produced by the new identified gene variants (qualitative and quantitative) and its effect on the platelet production by megakaryocytes in culture.

SECONDARY OUTCOMES:
Description of the phenotype of these new CT entities | 6 months
  Gathering information on a potentially associated clinical syndrome by a medical questionnaire reporting any organ dysfunction or pathology (renal impairment, deafness, malignancy, …) and collection of data of the blood cells counts. Blood cells counts will be compared to normal controls and data of the medical questionnaire will be compared between affected patients, in the aim to highlight the potential implication of the new gene variants in haematological or non haematological diseases.
Search of a potentially platelet dysfunction | 6 months
  Platelet function study by specialized techniques : activation and aggregation of cells (velocity, rate) in the presence of different platelet activators (ADP, collagen, thrombin) measured with aggregometer and flow immunocytometry, secretion measured with ELISA kits for specific platelet-secreted molecules and with flow immunocytometry, cell adhesion measured with optic and electronic microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Françoise Hurtaud-Roux, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (2):
- France (2):
  - Resource and Competence Center for Constitutional Hemorrhagic Diseases (CRCMHC), University Hospital Robert Debré, Paris
  - Resource and Competence Center for Constitutional Hemorrhagic Diseases (CRCMHC), University Hospital Pontchaillou, Rennes

REFERENCES:
- [Background] Vincenot A, Saultier P, Kunishima S, Poggi M, Hurtaud-Roux MF, Roussel A, Actn Study Coinvestigators, Schlegel N, Alessi MC. Novel ACTN1 variants in cases of thrombocytopenia. Hum Mutat. 2019 Dec;40(12):2258-2269. doi: 10.1002/humu.23840. Epub 2019 Nov 6. PMID 31237726
- [Background] Boutroux H, David B, Gueguen P, Frange P, Vincenot A, Leverger G, Favier R. ACTN1-related Macrothrombocytopenia: A Novel Entity in the Progressing Field of Pediatric Thrombocytopenia. J Pediatr Hematol Oncol. 2017 Nov;39(8):e515-e518. doi: 10.1097/MPH.0000000000000885. PMID 28562514
- [Background] Guillet B, Bayart S, Pillois X, Nurden P, Caen JP, Nurden AT. A Glanzmann thrombasthenia family associated with a TUBB1-related macrothrombocytopenia. J Thromb Haemost. 2019 Dec;17(12):2211-2215. doi: 10.1111/jth.14622. Epub 2019 Sep 29. PMID 31565851
- [Background] Balduini CL, Melazzini F, Pecci A. Inherited thrombocytopenias-recent advances in clinical and molecular aspects. Platelets. 2017 Jan;28(1):3-13. doi: 10.3109/09537104.2016.1171835. Epub 2016 May 9. PMID 27161842
- See also: Website of the Inserm U1140 laboratory "Innovative Therapeutics in Hemostasis" — http://www.ithem.fr/
- See also: Website of the rare diseases health chain "Mhemo" (meaning haemorrhagic diseases), which includes the CRCMHC — https://mhemo.fr/